CLINICAL TRIAL: NCT01998425
Title: Circulating Fibrocytes in Non-small Cell Lung Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB100-2929B-FibLC-CGMH
Record Dates: First submitted 2013-11-13; First posted 2013-11-28 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2013-10

CONDITIONS: NSCLC
Keywords: circulating fibrocytes; fibrocyte; NSCLC; treatment response; survival; stage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-small cell lung cancer: The cohort data of patients with NSCLC will follow up from diagnosis, treatment response and final survival. Fibrocytes will be checked on the date of diagnsis (before treatment), re-staing (3months after treatment) and disease progression.

SUMMARY:
The investigators will collect fibrocytes (CD45+Col-1+) in patients with non-small cell lung cancer (NSCLC). The investigators hypothesize that patients with NSCLC experience expansion of immunosuppressive fibrocytes, which are predicted to augment tumor growth by mediating immune escape in NSCLC patients.

DETAILED DESCRIPTION:
Fibrocytes have been described in both mice and humans, where they bear a hematopoietic progenitor phenotype (CD45+Col-1+). Fibrocytes have previously been described in murine cancer, implicated as mediators of tumor immune escape. In this study, the investigators will collect fibrocytes including CD45+Col-1+ expression. The cells express indoleamine oxidase, which is primarily responsible for their immunosuppressive properties. The investigators hypothesize that patients with non-small cell lung cancer experience expansion of immunosuppressive fibrocytes, which are predicted to augment tumor growth by mediating immune escape in non-small cell lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC).

Exclusion Criteria:

* Combination of other malignancy.
* Age less than 20 years (not include 20 years).
* Pregnancy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed non-small cell lung cancer (NSCLC) will be enrolled and evaluated from 2013 to 2016. Disease in all cases was staged with computed tomography (CT) of the chest, breast (if resectable) and positron emission tomography (PET, if resectable) within 3 months before enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-02 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
treatment response of participants by RECIST. | 18 months
  Correlation of circulating fibrocytes and treatment (chemotherapy, surgery, target treatment) response of patients with NSCLC.

SECONDARY OUTCOMES:
Survival of participants. | 24 months
  Correlation of circulating fibrocytes and survival (progression free survival, disease free survival and overall survival) of patients with NSCLC.

OTHER OUTCOMES:
Staging status of patients with NSCLC. | 18 months
  Correlation of circulating fibrocytes and stage of patients with NSCLC.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital, Linkou District
  - Chang Gung Memoral Hospital, Taoyuan District

REFERENCES:
- [Background] Weng CM, Chen BC, Wang CH, Feng PH, Lee MJ, Huang CD, Kuo HP, Lin CH. The endothelin A receptor mediates fibrocyte differentiation in chronic obstructive asthma. The involvement of connective tissue growth factor. Am J Respir Crit Care Med. 2013 Aug 1;188(3):298-308. doi: 10.1164/rccm.201301-0132OC. PMID 23795584
- [Background] Wang CH, Huang CD, Lin HC, Huang TT, Lee KY, Lo YL, Lin SM, Chung KF, Kuo HP. Increased activation of fibrocytes in patients with chronic obstructive asthma through an epidermal growth factor receptor-dependent pathway. J Allergy Clin Immunol. 2012 May;129(5):1367-76. doi: 10.1016/j.jaci.2012.01.038. Epub 2012 Feb 9. PMID 22325070
- [Background] Wang CH, Huang CD, Lin HC, Lee KY, Lin SM, Liu CY, Huang KH, Ko YS, Chung KF, Kuo HP. Increased circulating fibrocytes in asthma with chronic airflow obstruction. Am J Respir Crit Care Med. 2008 Sep 15;178(6):583-91. doi: 10.1164/rccm.200710-1557OC. Epub 2008 Jun 26. PMID 18583572
- [Background] Chung FT, Lee KY, Wang CW, Heh CC, Chan YF, Chen HW, Kuo CH, Feng PH, Lin TY, Wang CH, Chou CL, Chen HC, Lin SM, Kuo HP. Tumor-associated macrophages correlate with response to epidermal growth factor receptor-tyrosine kinase inhibitors in advanced non-small cell lung cancer. Int J Cancer. 2012 Aug 1;131(3):E227-35. doi: 10.1002/ijc.27403. Epub 2012 Jan 11. PMID 22174092
- [Background] Zhang H, Maric I, DiPrima MJ, Khan J, Orentas RJ, Kaplan RN, Mackall CL. Fibrocytes represent a novel MDSC subset circulating in patients with metastatic cancer. Blood. 2013 Aug 15;122(7):1105-13. doi: 10.1182/blood-2012-08-449413. Epub 2013 Jun 11. PMID 23757729
- [Background] Feng PH, Lee KY, Chang YL, Chan YF, Kuo LW, Lin TY, Chung FT, Kuo CS, Yu CT, Lin SM, Wang CH, Chou CL, Huang CD, Kuo HP. CD14(+)S100A9(+) monocytic myeloid-derived suppressor cells and their clinical relevance in non-small cell lung cancer. Am J Respir Crit Care Med. 2012 Nov 15;186(10):1025-36. doi: 10.1164/rccm.201204-0636OC. Epub 2012 Sep 6. PMID 22955317
- [Background] Liu CY, Wang YM, Wang CL, Feng PH, Ko HW, Liu YH, Wu YC, Chu Y, Chung FT, Kuo CH, Lee KY, Lin SM, Lin HC, Wang CH, Yu CT, Kuo HP. Population alterations of L-arginase- and inducible nitric oxide synthase-expressed CD11b+/CD14(-)/CD15+/CD33+ myeloid-derived suppressor cells and CD8+ T lymphocytes in patients with advanced-stage non-small cell lung cancer. J Cancer Res Clin Oncol. 2010 Jan;136(1):35-45. doi: 10.1007/s00432-009-0634-0. PMID 19572148